CLINICAL TRIAL: NCT04102332
Title: Evaluation of a Safe Infusion Device in Reducing Occupational Exposure of Nurses to Antineoplastic Drugs: a Comparative Prospective Study. CONTAMOINS-1
Brief Title: Safe Infusion Device in Reducing Occupational Exposure of Nurses
Acronym: CONTAMOINS-1
Status: Completed | Type: Observational
Sponsor: Institut de Cancérologie de la Loire (Other)
Collaborators: Centre Hospitalier Lyon Sud (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-PH1; IRBN522017/CHUSTE (Other: Comité d'Ethique du CHU de Saint-Etienne)
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Cancer
Keywords: Antineoplastic Agents; Cancer; Drug administration; Infusion device; Occupational Exposure; Nursing
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before arm: usual infusion practices (neutral solvent-purged infusers)
- After arm: Safe Infusion Device
  Interventions: Device: Safe Infusion Device

INTERVENTIONS:
Device: Safe Infusion Device — Safe infusion device is a different method than usual infusion practices (neutral solvent-purged infusers)
  Groups: After arm

SUMMARY:
Monocentric comparative before / after study to evaluate the efficacy of Safe Infusion Devices (SIDs) in reducing drug exposure to nurses compared to usual perfusion practices.

DETAILED DESCRIPTION:
Despite the decreasing of environmental contamination throughout the anticancer drug circuit, the administration of chemotherapies remains at risk of occupational exposure for nurses. Many medical devices aim at securing administration, but none have been scientifically evaluated to verify the actual improvement.

A monocentric comparative before / after study was carried out in an oncology day hospital in order to evaluate the efficacy of Safe Infusion Devices in reducing drug exposure compared to usual perfusion practices (neutral solvent-purged infusers). The rate of nurses' gloves contamination was estimated. The eligible protocols must contain at least one disconnection step and one of the 10 drugs screened. To avoid false negatives, each sample of gloves was contaminated with a drop of topotecan. Association between contamination and other variables was investigated using a multivariate regression analysis.

The usual practice leaded to a rate of 58.3% of contaminated samples while Safe Infusion Devices to a rate of 15%: Safe Infusion Devices reduced the risk of gloves contamination by 84% in multivariate analysis (Odds ratio=0.16; 95% confidence interval=0.05-0.47; p<0.001). Topotecan was identified within 100% of the samples. Only one case of cross-contamination has occurred.

Despite the current practice of using neutral solvent-purged infusers, the occupational exposure remains high for nurses and Safe Infusion Devices significantly reduced this risk of exposure. However, glove contamination is only a surrogate endpoint. The results confirmed that the disconnection of empty bags resulted in occupational exposure. Except a contamination due to the leakage of a bag, no cross-contamination was detected. This validated the environmental quality of the cytotoxic drug circuit. Safe Infusion Devices were highly effective but did not completely eliminate exposure.

ELIGIBILITY:
Inclusion Criteria:

* Protocols which contained at least one of the 10 drugs of the dosing assay
* Protocols with at least one disconnection step.
* Given the large number of eligible protocols, we favored those with the most concentrated products (CPM, PMX) to maximize the chance of detecting contamination and also to extend inclusions over a longer period.

Exclusion Criteria:

- Drugs administrated with syringes (intravenously or subcutaneously) were not included because of the absence of impact of the SIDs on these modalities of administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nurses that have to manipulate drugs for chemotherapies and that meet risks of contamination were asked to paritipate at the study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-08 (Actual)

PRIMARY OUTCOMES:
Rate of contamination of nurses' gloves with cytotoxic products | day 1
  The statistical unit consists of a sample taken from all the gloves used for the administration of a daily course. The dosing assay allowed to identify a panel of 10 cytotoxic drugs (HPLC MS/MS).

SECONDARY OUTCOMES:
Quantitative contamination of nurses' gloves with cytotoxic products | day 1
  The dosing assay allowed to identify a panel of 10 cytotoxic drugs (HPLC MS/MS).
Costs | day 1
  For each daily course performed in 2017 requiring the intravenous route, the necessary devices were estimated according to the two strategies
Manufacturing time | day 1
  The manufacturing time was defined as the time elapsed between the time of passage in the cleanroom and the end of manufacturing of the first drug of the course.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez, France

IPD SHARING:
Plan to Share IPD: No